CLINICAL TRIAL: NCT06694272
Title: Functional and Anatomical Visual Investigations in Patients With Early Forms of Age-related Macular Degeneration
Acronym: NOGA1
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SBN_2024_7
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subjects with early or intermediate AMD (normal visual acuity): At inclusion patients will have :
  * Measurements of subjective refraction, visual acuity, intraocular pressure, slit-lamp examination
  * Measurement of low-luminance visual acuity
  * Measurement of low-light contrast sensitivity
  * Photometric (> 30 cd/m² > 10 min) and scotopic (DA > 20 min) microperimetry
  * Multifocal electroretinogram
  * Imaging using fundus photography, OCT, OCT-A, adaptive optics and autofluorescence
  * Venous blood sampling (48 mL)
  After 4 years of follow-up, AMD evolution will be assessed with :
  * Measurements of subjective refraction, visual acuity, intraocular pressure, slit-lamp examination
  * Imaging by fundus photography, OCT, OCT-A, and autofluorescence

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of visual impairment in industrialized countries. Anatomical examination findings at the early and intermediate stages of AMD are not sufficient to determine any functional alterations at these stages (e.g., alterations in microperimetry, multifocal electroretinogram (mfERG) and contrast sensitivity). Identifying early functional markers of the disease is a necessary first step in the development and clinical validation of treatments to slow progression to advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Corrected visual acuity 10/10 in each eye
* Presence of retinal alteration(s) compatible with early (presence of macular drusen < 125 μm) or intermediate (macular drusen > 125 μm or pigmentary abnormalities) AMD in at least one of the two eyes :

  * Conventional "soft" or "hard" drusen
  * Cuticular drusen
  * Reticulated pseudo-drusen

Exclusion Criteria:

* Presence of geographic atrophy, even incipient, in one or both eyes
* Presence of patent or latent neovascularization visible on OCT b-scan or OCT-A in one or both eyes
* Compatibility of retinal signs with a "probable" differential diagnosis (bestrophinopathies, familial drusen, fundus flavimaculatus, fundus albipunctatus, hypovitaminosis A) in one or both eyes.
* Oculomotor pathology that may prevent proper performance of functional tests: nystagmus, oculomotor paralysis, in one or both eyes
* Neurological/neurodegenerative pathology that may prevent adequate performance of functional tests: advanced Parkinsonian syndromes, Benson's disease, Alzheimer's disease with visuomotor apraxia
* Other ophthalmological pathology that may affect anatomical and functional measurements: hypertonia / glaucoma or other optic neuropathy, media disorder causing reduced visual acuity, refraction < -6.00D or > +6.00D
* Other medical conditions preventing examinations or imaging (tremors, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with early or intermediate AMD (normal visual acuity)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
AMD evolution at 4 years | Year 4
  AMD is considered to have progressed if, after 4 years, the patient has developed an advanced form of the disease. The onset of an advanced form is defined by the appearance of macular neovascularization (of any type), visible on fundus or OCT/OCT-A, or by the appearance of macular atrophy visible on fundus, autofluorescence or OCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France